CLINICAL TRIAL: NCT06558149
Title: The Effect of Nociception Level (NOL) Monitoring on Intraoperative Opioid Consumption in Hip Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hadi Ufuk Yörükoğlu, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAD-DD- 01
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Post Operative Pain; Opioid Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analgesic use according to hemodynamics patients to be treated (Active Comparator): Procedure/Surgery: Pericapsular nerve group block(PENG) Before the general anesthesia induction, Peng block will be performed between the psoas tendon and the ilium with 0.25% bupivacaine (20 mL) using ultrasound and will be adjusting opioid infusion rate according to hemodinamic parameters
  Interventions: Procedure: Those whose opioids were adjusted according to hemodynamic parameters
- Patients who will use analgesics according to NOL monitoring (Active Comparator): Procedure/Surgery: Pericapsular nerve group block(PENG) Before the general anesthesia induction, Peng block will be performed between the psoas tendon and the ilium with 0.25% bupivacaine (20 mL) using ultrasound and will be adjusting opioid infusion rate according to NOL monitoring.
  Interventions: Procedure: Those whose opioids were adjusted according to NOL monitoring

INTERVENTIONS:
Procedure: Those whose opioids were adjusted according to hemodynamic parameters — Patient who will be adjusted according to hemodynamic parameter
  Arms: Analgesic use according to hemodynamics patients to be treated
Procedure: Those whose opioids were adjusted according to NOL monitoring — Patient who will be adjusted according to NOL monitoring
  Arms: Patients who will use analgesics according to NOL monitoring

SUMMARY:
Hip surgeries are one of the most painful surgical operations, and inadequate pain management increases postoperative morbidity and mortality.The incidence of chronic pain after hip surgery is quite high, at 11-40%.For this reason, hip surgeries are complex and specialized surgeries in terms of pain management.According to the surgical procedures pioneered by the European Society of Regional Anesthesia, Pericapsular nerve block (PENG) block is among the recommendations with a high level of evidence for hip surgery in the multimodal analgesia steps guide.In the literature, there are studies comparing the postoperative analgesic effectiveness of PENG block in hip surgeries, but the results are contradictory.In addition, intraoperative pain monitoring was not used in these studies, instead intraoperative analgesia management was provided according to hemodynamic parameters, which may not be objective.Opioid infusion is used in analgesia management during the intraoperative period.While not providing effective analgesia due to insufficient opioid use will have effects, excessive opioid use also has many side effects.Therefore, it would not be correct to administer the same dose of opioid infusion to every patient. As seen in the data in the literature and in daily practice, hemodynamic parameters (such as heart rate, blood pressure) are used for pain monitoring of the patient under general anesthesia, and these parameters may change depending on many other factors.Although some devices that aim to provide pain monitoring by evaluating the effects of pain on the sympathetic system are available on the market, their usage areas have remained limited since their reliability has not been fully demonstrated. Nociception level index (NoL) monitoring provides effective monitoring as it evaluates each patient separately using different parameters (heart rate, heart rate variability, photo-plethysmographic waveform amplitude, skin conductance level, number of skin conductance fluctuations and their time derivatives).While planning this study, İnvestigators aimed to use NoL monitoring in hip surgery, where postoperative pain management is quite challenging and important, as it provides objective and personalized pain management in patients under general anesthesia.When other studies in the literature are examined, the effects of regional techniques have been compared only in the postoperative period.Its effects in the intraoperative period have not been evaluated on a patient basis, and the opioid infusion rate has been adjusted with hemodynamic findings, which are affected by many parameters such as bleeding and drug use.In this study, İnvestigators aim to compare the effects of intraoperative pain monitoring and personalized analgesia treatment and the regional technique both in the intraoperative period and in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) physical status classification I-IV patients who are planned to undergo hip surgery

Exclusion Criteria:

* Allergies to study medications
* serious renal, pulmonary, liver and endocrine diseases
* have a history of chronic pain
* Those with a history of bleeding diathesis
* Those with increased intracranial pressure
* Those with severe mitral and/or aortic stenosis
* patients with psychiatric diseases and communication difficulties

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Remifentanil consumption | Intraoperative
  Total amount of remifentanil used during the surgery (mg)
NRS Scores | Postoperative 1st, 6th, 12th and 24th hours
  Numeric Rating Scale scores, between 0-10 (0= no pain, 10=worst pain imaginable)
Morphine consumption | Postoperative 1st, 6th, 12th and 24th hours
  Amount of morphine in the postoperative period (mg)

SECONDARY OUTCOMES:
Rescue analgesic | Postoperative 1st, 6th, 12th and 24th hours
  The use of rescue analgesic
Nausea and vomiting | Postoperative 1st, 6th, 12th and 24th hours
  If the patient had nausea or vomiting, it will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hadi Ufuk Yörükoğlu, Principal Investigator — Kocaeli University, Department of Anesthesiology and Reanimation

IPD SHARING:
Plan to Share IPD: No